CLINICAL TRIAL: NCT04275076
Title: Holmium Laser Enucleation of the Prostate Versus Bipolar Transurethral Enucleation of the Prostate in Management of Benign Prostatic Hyperplasia A Randomized Controlled Trial
Brief Title: HoLEP Vs BPEP for Large Prostatic Adenoma
Acronym: enucleation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahmed Maher Gamil Ahmed Higazy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Maher Gamil Ahmed Higazy, assistant lecturer of urology/ Specialist, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWA000017585.
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: patients, data collector, and the statistician all were blinded to the type of intervention that was used in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium laser enucleation of the prostate (Experimental): Holmium laser enucleation of the prostate
  Interventions: Procedure: Holmium laser enucleation of the prostate versus bipolar transurethral enucleation of the prostate in management of benign prostatic hyperplasia
- bipolar transurethral enucleation of the prostate (Experimental): bipolar transurethral enucleation of the prostate
  Interventions: Procedure: Holmium laser enucleation of the prostate versus bipolar transurethral enucleation of the prostate in management of benign prostatic hyperplasia

INTERVENTIONS:
Procedure: Holmium laser enucleation of the prostate versus bipolar transurethral enucleation of the prostate in management of benign prostatic hyperplasia — comparison between 2 energy sources of enucleation in management of benign prostatic hyperplasia, holmium laser versus bipolar energy source in trans-urethral enucleation of the prostate

SUMMARY:
Benign prostatic hyperplasia (BPH) is one of the most common urinary disorders in elderly males. The symptoms of BPH include impaired physiological and functional well-being, which interferes with daily living.

At present, transurethral resection of the prostate (TURP) is the standard surgical treatment. However, the high rate of complications associated with TURP is a major drawback of this procedure.

Holmium laser enucleation of the prostate (HoLEP) was proven to be an effective surgical treatment for BPH with no prostate size limitation with adequate hemostasis, bipolar enucleation of the prostate (BPEP) has been introduced as an alternative energy source with a promising outcome with equal safety and efficacy

DETAILED DESCRIPTION:
Enlarged prostate represents the most common cause of lower urinary tract symptoms (LUTS) in elderly men including irritative, obstructive urinary symptoms or even urinary retention that significantly affects the quality life (QoL).

Transurethral resection of the prostate (TURP) represents the standard surgical technique for the management of benign prostatic hyperplasia (BPH) with a prostate size less than 80 ml. However, considerable morbidities are associated with larger sizes.

Endoscopic enucleation of the prostate (EEP) has been recognized as a treatment option for large prostatic adenomas, since first described by Hiraoka et.al, in 1986, it started to gain popularity despite the long learning curve. Many studies have evaluated its efficacy against the gold standard open prostatectomy in large prostate size more than 80ml and showed its safety and efficacy.

EEP represents an anatomical surgical technique resembling a surgeon's finger in open prostatectomy where any energy source that provides adequate haemostasis could be used. Many studies concluded that EEP relies on the surgeon's skills rather than the energy source itself. Holmium laser enucleation of the prostate (HoLEP) was first described by Gilling in 1998 and was proven to be effective with no prostate size limitation with adequate haemostasis, recently it has been approved as a standard treatment for large prostatic adenoma, bipolar enucleation of the prostate (BPEP) has been introduced as an alternative energy source with a promising outcome with equal safety and efficacy.

Few studies evaluated both techniques, one study was done by Shoma et al. showing no statistical difference regarding safety and efficacy between both techniques, another study conducted by Enikeev et al. reported earlier recovery and catheter removal with HoLEP compared to BPEP. However, cost-effectiveness was never been evaluated before between both techniques especially in developing countries.

With such scarce information, the investigators aimed through this study to compare these two energy sources in the enucleation procedure of the prostate in terms of safety, efficacy, and cost-effectiveness in the management of BPH in large prostatic adenoma more than 80 ml.

ELIGIBILITY:
Inclusion Criteria:

* Men who are fit for surgery and need a surgical resection of the prostate larger than 80 ml including:

  1. Bothersome LUTS with an IPSS score over 19
  2. Refractory hematuria
  3. Upper urinary tract affection
  4. Recurrent UTI secondary to prostatic enlargement
  5. Maximum uroflow rate (Qmax) below 10 ml/sec.
  6. bladder diverticula
  7. Urinary retention whether recurrent acute attacks with failure of medical treatment or chronic retention.

Exclusion Criteria:

* Patients with:

  1. Neurogenic bladder
  2. Previous prostate or urethral surgery
  3. Associated urethral stricture
  4. Prostate cancer diagnosed by TRUS biopsy
  5. Bladder stones,

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
operative time | 50-120 minutes
  form the beginning of endoscopic procedure till catheter insertion

SECONDARY OUTCOMES:
Enucleation efficacy of HoLEP | 12 months
  Mean Enucleation time (HoLEP) in minutes divided by Mean resected volume in grams
Enucleation efficacy of BEEP | 12 months
  Mean Enucleation time (BPEP) in minutes/ Mean resected volume in grams
Mean energy in (HoLEP) in joules | intra-operative finding
  Mean energy in (HoLEP) in joules
irrigation fluid | intra-operative finding
  Average Irrigation fluid used in each group in liters
catheter removal time | 1-7 days
  postoperative time till catheter removal
resected volume | intra-operative finding
  resected volume in grams
hemoglobin drop | intra-operative finding
  blood loss in dl/ml
conversion to other type of surgery | intra-operative finding
  conversion to other types of surgeries like TURP, open surgery, procedure abortion
Operative safety: | intra-operative finding
  capsular perforation, Yes/No
Operative safety: | intra-operative finding
  morcellation injury, Yes/No
early post operative complication | 1 month
  stress incontinence, Yes/No
early post operative complication | 1 month
  urinary tract infection, Yes/No
early post operative complication | 1 month
  urine retention, Yes/No
Postoperative efficacy: | 12 months
  IPSS: international prostate symptom score
Postoperative efficacy: | 12 months
  QoL: quality of life questionnaire
Postoperative efficacy: | 12 months
  Qmax (m/sec.) : peak flow rate
Postoperative efficacy: | 12 months
  PVRU (ml): post voiding residual urine
Postoperative efficacy: | 12 months
  PSA (ng/ml): prostatic specific antigen
Postoperative efficacy: | 12 months
  postoperative prostate volume assessment in grams
cost effectiveness | 12 months
  Running cost in Egyptian pounds of the following: irrigation fluid, hospital stay, fiber, loop, management of complication in each group
hospital stay | 1-7 days
  duration of postoperative hospital stay in days
Cost analysis | 1 year
  average running cost evaluation in both procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT04275076/Prot_SAP_000.pdf